CLINICAL TRIAL: NCT06790121
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of 3 Subcutaneous Dose Regimens of Lunsekimig (SAR443765) in Adult Participants With Moderate-to-severe Atopic Dermatitis
Brief Title: A Study to Investigate the Efficacy and Safety of Subcutaneous Lunsekimig (SAR443765) Compared With Placebo in Adult Participants With Moderate-to-severe Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRI18252; U1111-1299-1958 (Registry Identifier: ICTRP); 2024-511549-20 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Lunsekimig arm A (Experimental): Participants will receive subcutaneous injection of lunsekimig dosing regimen A.
  Interventions: Drug: Lunsekimig
- Placebo arm B (Placebo Comparator): Participants will receive subcutaneous injection of matching placebo.
  Interventions: Drug: Placebo
- Lunsekimig arm C (Experimental): Participants will receive subcutaneous injection of lunsekimig dosing regimen C.
  Interventions: Drug: Lunsekimig
- Placebo arm D (Placebo Comparator): Participants will receive subcutaneous injection of matching placebo.
  Interventions: Drug: Placebo
- Lunsekimig arm E (Experimental): Participants will receive subcutaneous injection of lunsekimig dosing regimen E.
  Interventions: Drug: Lunsekimig
- Placebo arm F (Placebo Comparator): Participants will receive subcutaneous injection of matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lunsekimig — Pharmaceutical form: Solution for injection in vial Route of administration: Subcutaneous injection
  Other Names: SAR443765
  Arms: Lunsekimig arm A; Lunsekimig arm C; Lunsekimig arm E
Drug: Placebo — Pharmaceutical form: Solution for injection in vial Route of administration: Subcutaneous injection
  Arms: Placebo arm B; Placebo arm D; Placebo arm F

SUMMARY:
This is a parallel, Phase 2b, randomized, double-blind, placebo-controlled, multicenter study to assess the efficacy, safety, and tolerability of lunsekimig monotherapy in adult participants (aged 18 to 80 years, inclusive) with moderate-to-severe atopic dermatitis (AD).

This study explores the efficacy and safety of 3 subcutaneous (SC) dose regimens of lunsekimig in adult participants with moderate-to-severe AD who have a documented history, within 6 months prior to baseline, of an inadequate response to topical treatments or for whom topical therapies are not advised. The study consists of 6 arms: 3 parallel dosing regimens and matching placebo arms. Additionally, participants have the option of engaging in a dense pharmacokinetic/pharmodynamic (PK/PD) sampling subgroup.

The study duration will be up to approximately 36 weeks, including up to 4 weeks of screening, 24 weeks of treatment period and an 8-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 80 years of age, inclusive, at the time of signing the informed consent.
* Diagnosis of Atopic Dermatitis (AD) as defined by the American Academy of Dermatology (AAD) clinical guidelines (2023) for 1 year or longer at baseline (Day 1)
* Documented history within 6 months prior to Screening Visit, of either inadequate response or inadvisability of topical treatments
* Eczema Area and Severity Index (EASI) score of 16 or higher (range, 0 to 72) at baseline (Day 1)
* Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) score of 3 or 4 at baseline visit (Day 1) (on the 0 to 4 vIGA-AD scale, a vIGA-AD score of 3 and 4 represents moderate and severe, respectively).
* AD involvement of 10% or more of Body Surface Are (BSA) at baseline (Day 1)
* Weekly average of daily Peak Pruritis-Numerical Rating (PP-NRS) score of ≥4 at baseline (Day 1)
* Must have applied a stable dose of topical bland emollient (simple moisturizer, no additives [eg, urea]) at least once daily for a minimum of 5 out of 7 consecutive days before baseline (Day 1).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Skin comorbidity that would adversely affect the ability to undertake AD assessments (eg, psoriasis, tinea corporis, and lupus erythematosus) according to the Investigator's judgment.
* Known history of, or suspected, significant current immunosuppression

NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Percent change in Eczema Area and Severity Index (EASI) score from baseline to Week 24 | From Baseline throughout the study, up to Week 24
  Eczema Area and Severity index is an Investigator-assessed validated tool used to measure the extent (area) and severity of atopic dermatitis (AD). Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.

SECONDARY OUTCOMES:
Proportion of participants achieving EASI-75 at Week 24 | From Baseline throughout the study, up to Week 24
  EASI 75 is defined by reduction of EASI score by ≥75% from baseline
Proportion of participants with a Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) score of 0 (clear) or 1 (almost clear) and a reduction from Baseline of ≥2 points at Week 24 | From Baseline throughout the study, up to Week 24
  The Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) score is a 5-point scale used to determine severity of AD and clinical response to treatment, ranging from 0 (clear) to 4 (severe).
Proportion of participants with reduction (improvement) of ≥4 in the weekly average of daily Peak Pruritis-Numerical Rating Scale (PP-NRS) score from Baseline to Week 24 | From Baseline throughout the study, up to Week 24
  The Peak Pruritis-Numerical Rating Scale (PP-NRS) is a validated single-item patient-reported outcome (PRO) to assess worst itch intensity on a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Absolute change from Baseline in EASI score at Week 24 | From Baseline throughout the study, up to Week 24
  Eczema Area and Severity index is an Investigator-assessed validated tool used to measure the extent (area) and severity of atopic dermatitis (AD). Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Percent change from Baseline in EASI score throughout the study | From Baseline throughout the study, up to Week 24
  Eczema Area and Severity index is an Investigator-assessed validated tool used to measure the extent (area) and severity of atopic dermatitis (AD). Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Proportion of participants with a vIGA-AD score of 0 (clear) or 1 (almost clear) at Week 24 | From Baseline throughout the study, up to Week 24
  The Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) score is a 5-point scale used to determine severity of AD and clinical response to treatment, ranging from 0 (clear) to 4 (severe).
Proportion of participants with a response of vIGA-AD 0 or 1 and a reduction from Baseline of ≥2 points throughout the study | From Baseline throughout the study, up to Week 24
  The Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) score is a 5-point scale used to determine severity of AD and clinical response to treatment, ranging from 0 (clear) to 4 (severe).
Percent change in the weekly average of daily PPNRS scores from Baseline to Week 24 | From Baseline throughout tje study, up to Week 24
  The Peak Pruritis-Numerical Rating Scale (PP-NRS) is a validated single-item patient-reported outcome (PRO) to assess worst itch intensity on a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Percent change in the weekly average of daily sleep disturbance NRS score from Baseline to Week 24 | From Baseline throughout the study, up to Week 24
  The Sleep Disturbance-Numerical Rating Scale (SD-NRS) is a validated single item 0-10 numerical rating scale assessing sleep disturbance associated with AD, with 0 being 'no sleep loss related to the symptoms of AD' and 10 being 'I did not sleep at all' due to the symptoms of AD.
Percent change in the weekly average of daily skin pain NRS score from Baseline to Week 24 | From Baseline throughout the study, up to Week 24
  The Skin Pain-NRS is a whole number scale ranging from 0 to 10 with a 24-hour recall period, with 0 = no pain and 10 = worst possible pain imaginable. The threshold for determining clinically meaningful change is ≥ 4-point change in the weekly average SP-NRS.
Change in percent Body Surface Area (BSA) affected by Atopic Dermatitis from Baseline to Week 24. | From Baseline throughout the study, up to Week 24
  The BSA affected by AD will be assessed in 4 body regions: head/neck, trunk (including the genitals), upper extremities, and lower extremities (including the buttocks). Each body region should be evaluated from 0 to 100%. The percentage of the affected area will be multiplied by the proportion of that body region to the whole body.
Proportion of participants achieving EASI-50 at Week 24 | From Baseline throughout the study, up to Week 24
  EASI-50 is defined by reduction of EASI score by ≥50% from baseline.
Proportion of participants achieving EASI-90 at Week 24 | From Baseline throughout the study, up to Week 24
  EASI-90 is defined by reduction of EASI score by ≥90% from baseline.
Proportion of participants with improvement (reduction) of ≥4 points in the weekly average of daily PP NRS scores from Baseline throughout the study | From Baseline throughout the study, up to Week 24
  The Peak Pruritis-Numerical Rating Scale (PP-NRS) is a validated single-item patient-reported outcome (PRO) to assess worst itch intensity on a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Proportion of participants with improvement (reduction) of ≥4 points in the weekly average of daily SD-NRS scores from Baseline to Week 24, in participants with a baseline weekly average of daily SD-NRS scores of ≥4 points | From Baseline throughout the study, up to Week 24
  The Sleep Disturbance-Numerical Rating Scale (SD-NRS) is a validated single item 0-10 numerical rating scale assessing sleep disturbance associated with AD, with 0 being 'no sleep loss related to the symptoms of AD' and 10 being 'I did not sleep at all' due to the symptoms of AD.
Proportion of participants with improvement (reduction) of ≥4 points in the weekly average of daily Skin Pain NRS scores from Baseline to Week 24, in participants with a baseline weekly average of daily Skin Pain NRS scores of ≥4 points | From Baseline throughout the study, up to Week 24
  The Skin Pain--Numerical Rating Scale (SP-NRS) is a whole number scale ranging from 0 to 10 with a 24-hour recall period, with 0 = no pain and 10 = worst possible pain imaginable. The threshold for determining clinically meaningful change is ≥ 4-point change in the weekly average SP-NRS.
Percent change in Scoring of Atopic Dermatitis (SCORAD) Index from Baseline to Week 24 | From Baseline throughout the study, up to Week 24
  The Scoring of Atopic Dermatitis (SCORAD) Index is a validated clinical tool that was developed to standardize the evaluation of the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Proportion of participants with an improvement of ≥4 points in Dermatology Life Quality Index (DLQI) score from Baseline to Week 24 and throughout the study | From Baseline throughout the study, up to Week 24
  The Dermatology Life Quality Index (DLQI) is a 10-item dermatology specific health-related quality of life (HRQoL) questionnaire. The total score is correlated to the detrimental effect of AD on QoL and ranges from 0 to 30, with a higher score indicating a poorer QoL.
Percent change in Dermatology Life Quality Index (DLQI) score from Baseline to Week 24 and throughout the study | From Baseline throughout the study, up to Week 24
  The Dermatology Life Quality Index (DLQI) is a 10-item dermatology specific health-related quality of life (HRQoL) questionnaire. The total score is correlated to the detrimental effect of AD on QoL and ranges from 0 to 30, with a higher score indicating a poorer QoL.
Percent change in Patient Oriented Eczema Measure (POEM) score from Baseline to Week 24 | From Baseline throughout the study, up to Week 24,
  The Scoring of Atopic Dermatitis (SCORAD) Index is a validated clinical tool that was developed to standardise the evaluation of the extent and severity of AD.
Percent change in Hospital Anxiety and Depression Scale (HADS) from Baseline to Week 24 | From Baseline throughout the study, up to to Week 24
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item patient-reported outcome (PRO) questionnaire used to assess states of anxiety and depression over the past week with two subscales. Each subscale (anxiety & depression) ranges 0-21. The total HADS score ranges 0-42 with higher score indicating a poorer state.
Incidence of Antidrug antibody (ADA) against lunsekimig up to end of study | From Baseline throughout the study, up to Week 32
Serum concentrations of lunsekimig throughout the study | From Baseline throughout the study, up to Week 32
Serum concentrations of lunsekimig in the pharmacokinetic/pharmacodynamics (PK/PD) subgroup throughout the study | From Baseline throughout the study, up to Week 32
Number of participants with treatment-emergent adverse events (TEAEs), including local reactions, adverse events of special interest (AESIs), and serious adverse events (SAEs) | From Baseline throughout the study, up to Week 32

CONTACTS AND LOCATIONS:
Locations (52):
- United States (23):
  - T. Joseph Raoof MD Inc-Site Number: 8400004, Encino, California
  - Integrative Skin Science and Research-Site Number: 8400002, Sacramento, California
  - Clinical Trials Research Institute-Site Number: 8400003, Thousand Oaks, California
  - Skin Care Research-Site Number: 8400013, Boca Raton, Florida
  - Driven Research LLC-Site Number: 8400020, Coral Gables, Florida
  - Revival Research Institute, LLC-Site Number: 8400021, Evans, Georgia
  - Treasure Valley Medical Research-Site Number: 8400026, Boise, Idaho
  - Southern Indiana Clinical Trials-Site Number: 8400024, New Albany, Indiana
  - Indiana Clinical Trials Center, P.C.-Site Number: 8400018, Plainfield, Indiana
  - Optima Research-Site Number: 8400019, Plainfield, Indiana
  - Options Research Group-Site Number: 8400012, West Lafayette, Indiana
  - DS Research - Kentucky-Site Number: 8400005, Louisville, Kentucky
  - Clinical Trials Management LLC-Site Number: 8400010, Covington, Louisiana
  - Beacon Clinical Research-Site Number: 8400006, Quincy, Massachusetts
  - Somerset Skin Centre-Site Number: 8400009, Troy, Michigan
  - Medisearch LLC-Site Number: 8400017, Saint Joseph, Missouri
  - Skin Cancer and Dermatology Institute-Site Number: 8400011, Reno, Nevada
  - Icahn School of Medicine at Mount Sinai-Site Number: 8400023, New York, New York
  - Red River Research Partners-Site Number: 8400008, Fargo, North Dakota
  - Health Concepts-Site Number: 8400025, Rapid City, South Dakota
  - DermResearch-Site Number: 8400014, Austin, Texas
  - Progressive Clinical Research-Site Number: 8400001, San Antonio, Texas
  - Burien US-WA 98168 Dermatology of Seattle and Bellevue-Site Number: 8400015, Burien, Washington
- Czechia (4):
  - Investigational Site Number: 0203003, Prague
  - Investigational Site Number: 0203001, Prague
  - Investigational Site Number: 0203004, Prague
  - Investigational Site Number: 0203002, Prague
- Japan (8):
  - Investigational Site Number: 3920005, Asahikawa-shi
  - Investigational Site Number: 3920003, Fukuoka
  - Investigational Site Number: 3920004, Kofu
  - Investigational Site Number: 3920002, Mibu
  - Investigational Site Number: 3920006, Nerima-ku
  - Investigational Site Number: 3920001, Ōta-ku
  - Investigational Site Number: 3920008, Tachikawa-shi
  - Investigational Site Number: 3920007, Yokohama
- Poland (17):
  - Investigational Site Number: 6160014, Bochnia
  - Investigational Site Number: 6160006, Bydgoszcz
  - Investigational Site Number: 6160010, Jelenia Góra
  - Investigational Site Number: 6160007, Katowice
  - Investigational Site Number: 6160003, Katowice
  - Investigational Site Number: 6160013, Lublin
  - Investigational Site Number: 6160001, Mikołów
  - Investigational Site Number: 6160011, Nowa Sól
  - Investigational Site Number: 6160015, Ostrowiec Swietokrzyskie
  - Investigational Site Number: 6160009, Poznan
  - Investigational Site Number: 6160012, Sosnowiec
  - Investigational Site Number: 6160004, Szczecin
  - Investigational Site Number: 6160017, Warsaw
  - Investigational Site Number: 6160018, Warsaw
  - Investigational Site Number: 6160002, Warsaw
  - Investigational Site Number: 6160005, Wroclaw
  - Investigational Site Number: 6160016, Łodź

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI18252 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26517&tenant=MT_SNY_9011